CLINICAL TRIAL: NCT02974504
Title: A Multicenter, Randomized, Double-blind, Active-contrelled, Parallel-group, Phase IV Clinical Trial to Investigate the Effect on Blood Glucose of Evogliptin After Oral Administration in Patiend With Type 2 Diabetes
Brief Title: Phase IV Clinical Trial to Investigate the Effect on Blood Glucose of Evogliptin in Patients With Type 2 Diabetes(EVERGREEN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1229_DM_IV
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- evogliptin (Experimental): evogliptin 5mg qd
  Interventions: Drug: evogliptin
- linagliptin (Active Comparator): linagliptin 5mg qd
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: evogliptin — evogliptin 5mg tablet qd + placebo tablet matching to linagliptin 5mg
  Arms: evogliptin
Drug: Linagliptin — linagliptin 5 mg tablet qd + placebo tablet matching to evogliptin 5mg
  Other Names: Tragenta
  Arms: linagliptin

SUMMARY:
A multi-center, randomized, double-blind, active-controlled, parallel group, phase IV clinical trial to investigate the effect on blood glucose of evogliptin after oral administration in patients with type 2 diabetes

DETAILED DESCRIPTION:
1. Evogliptin 5mg Group: Administration with Evogliptin 5mg for 0-24 weeks.
2. Liniagliptin 5mg Group: Administration with linagliptin 5mg for 0-12 weeks, and with Evogliptin 5mg for 13-24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subjects with 7.0%≤HbA1c≤10.0% at screening

  * Subjects untreated with oral hypoglycemic agents within 8 weeks prior to screening
* Subjects with 20kg/m2≤BMI≤40kg/m2 at screening

Exclusion Criteria:

* Subjects with fasting plasma glucose≥270mg/dL at screening
* Patients with type 1 diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* Subjects with history of myocardial infarction, cerebral infarction within 24 weeks prior to screening
* Subjects with ALT and AST 3 times or higher than upper normal range

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from baseline at 12 week
  unit: %

SECONDARY OUTCOMES:
fasting plasma glucose | Change from baseline at 12 week
  unit : mg/dL
HbA1c response rate | Change from baseline at 12 weeks
  unit: %

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology and Metabolism, Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No